CLINICAL TRIAL: NCT04024748
Title: Verification of Imaging System PCD-1000A
Status: Completed | Type: Observational
Sponsor: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: PCD-1000A
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2019-07

CONDITIONS: Cancer Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients already scheduled for a FDG test: Subjects will be selected from patients already scheduled for a routine FDG PET/CT test. Only adult patients, 40 years old or older, capable of providing their informed consent, will be selected. Any adult female patients that are pregnant and/or could become pregnant will be excluded. Twenty patients will be recruited.
  Interventions: Device: PET/CT imaging

INTERVENTIONS:
Device: PET/CT imaging — Subjects will be have a PET/CT scan with PCD-1000A following their scheduled routine PET/CT scan. There will be no additional administration of radiopharmaceutical for the study.

SUMMARY:
Scope Verification of technologies included in the PCD-1000A PET/CT imaging chain.

* Define and confirm all supported clinical protocols
* Evaluate performance

DETAILED DESCRIPTION:
The study aim is system verification and associated software. Clinical data and clinical feedback will be used for verification.

ELIGIBILITY:
Inclusion Criteria:

* Patients already scheduled for an FDG test at SDMI
* 40 years and older
* Capable of providing their informed consent

Exclusion Criteria:

* Patients not scheduled for an FDG test at SDMI
* 39 years or younger
* Adult female patients that are and/or could become pregnant
* Not capable of providing their informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Cancer Patients, 40 years or older, scheduled for a standard-of-care PET/CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Confirm that PCD-1000A PET/CT System is Effective for Its Intended Use | 3 months
  PCD-1000A PET/CT system's performance will be evaluated for oncology PET imaging on cancer patients to verify that the system performs as expected.
  • Verify that all supported clinical protocols from PET acquisition, reconstruction, to presentation (filtering) perform as expected. Images acquired by PCD-1000A PET/CT will be compared with images acquired during a standard-of-care PET/CT scan by a commercially available PET/CT system just prior to imaging with the PCD-1000A PET/CT System. Image quality evaluation will include assessment of uniformity of the liver, delineation of the lungs, presence of artifacts and using Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Steinberg Diagnostic Medical Imaging Centers, Henderson, Nevada, United States